CLINICAL TRIAL: NCT06149845
Title: Treatment Outcomes of Pulpotomy in Vital Primary Molars Diagnosed With Symptomatic Irreversible Pulpitis: An International Multi-centre Study
Brief Title: Pulpotomy in Vital Primary Molars Diagnosed With Symptomatic Irreversible Pulpitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qatar University (Other)
Collaborators: Primary Health Care Corporation, Qatar (Other Government); Jordan University of Science and Technology (Other); King Abdulaziz Hospital, Saudi Arabia (Unknown); Dubai Dental Hospital (Unknown); Cairo University (Other); Hamdan Bin Mohammed College of Dental Medicine (Unknown)
Responsible Party: Principal Investigator, Nebu Philip, Assistant Professor, Qatar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QU2713
Record Dates: First submitted 2023-11-18; First posted 2023-11-29 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Irreversible Pulpitis
Keywords: Pulpotomy

STUDY DESIGN:
Intervention Model Description: Longitudinal prospective single-arm cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pulpotomy (Experimental): Participants diagnosed with symptomatic irreversible pulpitis in vital primary molars will receive the pulpotomy treatment intervention
  Interventions: Procedure: Full Pulpotomy

INTERVENTIONS:
Procedure: Full Pulpotomy — Pulpotomy is a more conservative pulp treatment option where only the coronal pulp is removed and a medicament placement over the remnant radicular pulp after haemostasis is achieved.

SUMMARY:
This is a clinical trial to assess the treatment outcomes of pulpotomy in vital primary molars diagnosed with symptomatic irreversible pulpitis. Pulpotomy is a more conservative treatment option over the conventional pulpectomy treatment. Compared to pulpectomy, pulpotomy is a technically simpler procedure, less time consuming, easier for young patients to tolerate, and retains the proprioceptive sensation of the tooth - all important advantages when treating young children.

DETAILED DESCRIPTION:
Background: Pulpectomy continues to be the standard treatment recommendation for management of vital primary molars diagnosed with symptomatic irreversible pulpitis. The recent decade has seen a paradigm shift in the treatment concepts of how vital mature permanent molars diagnosed with irreversible pulpitis can be more conservatively managed using vital pulp therapy techniques like pulpotomy. However, despite emerging evidence indicating similarities between primary and permanent tooth pulp response to dental caries, there is limited research on whether pulpotomy can be similarly used as a definitive treatment modality for vital primary teeth diagnosed with irreversible pulpitis.

Aim: This study primarily aims to assess the clinical and radiographic treatment outcomes of full pulpotomy in vital primary molars diagnosed with symptomatic irreversible pulpitis.

Methods/Design: Healthy cooperative children, between 4-9 years of age, who have painful primary molars with symptoms typical of irreversible pulpitis will be recruited for the study from paediatric dental clinics located in eight countries (Qatar, Saudi Arabia, Kuwait, U.A.E, Jordan, Egypt, U.S.A, and Thailand). The primary outcome that will be assessed are the clinical success rates after one-year and two-years of the pulpotomy intervention. The secondary outcomes that will be assessed include: (i) immediate post-operative pain relief after 24 h and 7-days of the pulpotomy intervention; and (ii) radiographic success rates after one-year and two-years of the pulpotomy intervention. The influence of baseline pre-operative variables (age; gender; tooth type; site of caries; pre-operative furcal radiolucency; pre-operative pain intensity) and intra-operative factors (time taken to achieve haemostasis) on treatment outcomes will also be evaluated.

Discussion: This clinical trial seeks to provide evidence on whether pulpotomy can be used for the management of vital primary molars diagnosed with symptomatic irreversible pulpitis

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (ASA I and II) co-operative children (Frankl Scale + and ++) between the ages of four and nine years.
2. Participants have symptoms typical of irreversible pulpitis in one of the primary molars.
3. The pulp of the affected primary molar is vital.
4. Radicular pulp health is confirmed by attainment of radicular pulp haemostasis within 6 minutes of coronal pulp amputation.
5. The affected primary molars can be restored with full coverage crowns.
6. Any physiologic root resorption, if present, is less than ⅓ the root length

Exclusion Criteria:

1. Clinical examination of affected primary molar reveals signs of pulpal infection (e.g.

   pathologic tooth mobility, parulis/fistula, or soft tissue swelling)
2. Pre-operative periapical radiograph suggests presence of periapical radiolucency.
3. Pre-operative periapical radiograph suggests presence of furcal radiolucency more than ½ the furcation to periapical area.
4. Visual examination of pulp tissue after deroofing reveals signs of necrosis (e.g.

   avascular/minimally bleeding pulp tissue or yellowish necrotic areas/purulent exudate).
5. Signs of extensive radicular pulp inflammation.
6. Parents not willing to place full coverage crowns post-pulpotomy.
7. Clinical diagnosis of irreversible pulpitis between two teeth is not sharply defined.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Post-treatment clinical success | 6 months, 12 months, 24 months
  Clinical success will be determined at 6-, 12-, and 24-months based on the pulpotomy treated tooth meeting all the below criteria:
  * Treated tooth is not associated with any pain or discomfort
  * Treated tooth is not associated with tenderness on percussion or palpation
  * Treated tooth is not associated with any swelling, parulis, or fistula
  * Treated tooth is not associated with any pathological mobility

SECONDARY OUTCOMES:
Immediate post-treatment pain relief | 24 hours; 7 days
  Pain scores that will be recorded at 24-hours and 7-days post-treatment using a child friendly Visual Analogue Scale (VAS). This pain score will be used to evaluate pain reduction afforded by the pulpotomy treatment intervention.
Post-treatment radiographic success | 6 months, 12 months, 24 months
  Radiographic success will be determined at 6-, 12-, and 24-months based on the pulpotomy treated tooth meeting all the below criteria:
  * No signs of pathological internal/external root resorption or new furcal/periapical lesions on recall periapical radiographs
  * Complete radiographic healing or reduction/no change in size of any pre-treatment furcal rarefaction on recall periapical radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Nebu Philip, PhD, Principal Investigator — Qatar University
Locations (2):
- Qatar (2):
  - Phcc - Airport Center, Doha
  - PHCC- Leebaib Center, Doha

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Philip N, Kowash M, Bani-Hani T, Shahawy OE, Issa A, Mohamed H, Abdalla M, Jundi S, Albadri S, Duggal M, Nazzal H. Pulpotomy for treating primary molars with clinical symptoms indicative of irreversible pulpitis: A prospective single-arm pilot study. J Dent. 2025 Dec;163:106140. doi: 10.1016/j.jdent.2025.106140. Epub 2025 Sep 28. PMID 41027503